CLINICAL TRIAL: NCT05031325
Title: A Multicenter Randomized Controlled Trial to Evaluate the Efficacy of a Hemostatic Agent (PuraStat®) in Reducing Delayed Bleeding After Endoscopic Colorectal Submucosal Dissection
Brief Title: Efficacy of a Hemostatic Agent (PuraStat®) in Reducing Delayed Bleeding After Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mathieu Pioche (Other)
Responsible Party: Sponsor-Investigator, Mathieu Pioche, Principal Investagator, Medical Doctor, Société Française d'Endoscopie Digestive
Organization: Société Française d'Endoscopie Digestive (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFED 151
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Colo-rectal Cancer
Keywords: Resection; Colorectal lesions; bleeding; ESD
MeSH Terms: conditions — Colonic Neoplasms; Hemorrhage | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic submucosal dissection with Purastat (Experimental): To compare of the risk of bleeding after endoscopic submucosal dissection, after ESD, application of Purastat gel (not a drug but a device with CE mark) with a catheter of a gel on the resected area to cover the whole surface of mucosal resection.
  Interventions: Device: Endoscopic submucosal dissection with Purastat
- Comparative arm without Purastat (No Intervention): After endoscopic submucosal dissection (ESD) and hemostasis, if the patient is randomized in the comparative group, no gel will be applied on the resected area that will remain like this without intervention (common practice)

INTERVENTIONS:
Device: Endoscopic submucosal dissection with Purastat — Purastat (peptidic gel) application
  Arms: Endoscopic submucosal dissection with Purastat

SUMMARY:
The problem of delayed bleeding after endoscopic resection is becoming important due to the growing number of indications for anti-aggregation or anticoagulant treatment for cardiovascular reasons in the aging populations. Previous studies have shown that in patients at high risk of bleeding, the use of (PuraStat®), a simple and easily applicable solution, decreases the rate of delayed bleeding by promoting wound healing. Various preventive treatments, such as the prophylactic use of clips, have been tried to prevent the occurrence of delayed bleeding, but to date, no treatment has clearly shown its effectiveness. In addition, preventive hemostasis with clips is difficult and costly. The main objective is to compare the efficacy of PuraStat® to the standard treatment in reducing delayed bleeding after colorectal ESD in patients at high risk of delayed bleeding. The secondary objectives are to compare the same two strategies in terms of effectiveness and side effects. The primary outcome measure is the percentage of delayed bleeding at 30 days after surgery (ESD).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18 years or older
* Patient with a validated indication for colonoscopy for colorectal lesions
* Patients with a single colorectal lesion to be resected by ESD according to European recommendations.
* Patients with a colorectal neoplastic lesion (≥3 cm)
* Patients taking anticoagulants (acetylsalicylic acid >300 mg/day) or antiplatelet agents (clopidogrel, prasugrel, ticagrelor, clopidogrel) and managed according to European recommendations for ESD (including patients who may require heparin replacement)
* Written consent signed after clear, fair, and understood information.
* Patients with social security coverage.

Exclusion Criteria:

* Patients who may have an allergic reaction to the substances of PuraStat®.
* Patients with severe fibrosis
* Patients with a history of familial colorectal polyposis (familial adenomatous, Lynch syndrome, Peutz-Jeghers syndrome)
* Patients with a score ASA greater than or equal to 4 or 5
* Patients with a platelet count of 50,000/mm3
* Patients with acquired (non-medicated) or inherited bleeding disorders
* Patients who are being treated with acetylsalicylic acid but whose treatment is discontinued at the time of the procedure (therapeutic window)
* Patients with advanced cancer or inflammatory bowel disease, including ulcerative colitis (with colonic involvement)
* Contraindication to general anesthesia
* Patients with a mental disorder, drug addiction, alcoholism, etc.
* Pregnant women or women wishing to become pregnant during the study
* Patients already participating or scheduled to participate in other clinical trials
* Lesion that has been previously resected by mucosectomy
* Patient with an initial metastatic lesion prior to colonoscopy.
* Patient unable to give personal consent
* Lack of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of delayed bleeding after surgery (ESD) | through study completion, an average of 2 year
  Percentage of delayed bleeding is expressed primarily by the number of patients with at least one unplanned colorectal endoscopy occurring within 30 days of surgery (ESD)

SECONDARY OUTCOMES:
Rate of emergency endoscopy use by risk factors for secondary bleeding | through study completion, an average of 2 year
  Number of patients with at least one unplanned colorectal endoscopy by factors for secondary bleeding occurring within 30 days of ESD.
Rate of emergency endoscopic hemostasis use by risk factors for secondary bleeding | through study completion, an average of 2 year
  Number of patients requiring hemostasis, unplanned occurring within 30 days of ESD.
Rate of cases requiring transfusion related to post-ESD bleeding | through study completion, an average of 2 year
  Number of patients for whom at least one transfusion was ordered after the ESD
Rate of adverse events related to procedures (delayed perforation and stenosis) in each of the 2 arms | through study completion, an average of 2 year
  Number of patients with at least one delayed perforation or one symptomatic stenosis.
Rate and duration of hospitalizations | through study completion, an average of 2 year
  Number of hospitalizations and number of days of hospitalization per stay within 30 days after ESD
Tolerance of PuraStat | through study completion, an average of 2 year
  Number of patients with at least one irritation or thromboembolic accidents.
Evaluation of the gel application time on the resection area | During the intervention
  Time between introduction and removal of the PuraStat® catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France